CLINICAL TRIAL: NCT04746846
Title: SCH: Context-aware Freezing of Gait Mitigation in Real-world Setting
Status: Completed | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20020085; R01NS120560 (NIH)
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Vibration therapy (Experimental): 5-meter walk scenarios with vibration therapy
  Interventions: Device: UG motion sensor with PDVibe3

INTERVENTIONS:
Device: UG motion sensor with PDVibe3 — UG motion sensor (which detects FoG) on worn each ankle. PDVibe3 (which provides vibration) on worn each ankle

SUMMARY:
People with Parkinson's disease (PD) may experience a walking problem called freezing of gait (FoG) that can interfere with the person's ability to conduct daily activities. FoG has been described as feeling like one's feet are glued or stuck to the floor. Drug treatments for PD rarely improve FoG. Researchers have found that vibration therapy may help improve FoG. The purpose of this research study is to test the safety, tolerability, and effectiveness of using a wearable device (UG motion sensor, that is the size of a watch) that will recognize FoG and then send a signal to another small watch-like device (PDVibe3) to deliver a vibration stimuli to participant's feet. The researchers believe the vibration stimulus (which feels like a phone on vibration mode) will help reduce FoG in persons with PD. The study is open to people who have been diagnosed with Parkinson's disease, have FoG, and meet the study entry requirements.

The PDVibe3 is an investigational device, which means it has not been approved by the U.S. Food and Drug Administration (FDA). The UG motion sensor is also an investigational device.

DETAILED DESCRIPTION:
Usual care for PD involves taking medications to help with disease. In this study, participants will receive usual care. Participants will be asked to have taken their medication before they arrive, and to bring extra medicine with them should their next dose be due while they are at the study site.

Participants will be asked to walk on certain paths, and when the device detects a freeze in their gait, they will receive a dose of vibration to their feet. This vibration is felt differently by different people and it may feel very light or a little stronger (like a phone set to vibrate), or it may feel somewhere in between.

During the study, participants will be asked to do the following things:

1. Visit the research site at VCU, one time for the study
2. Complete a short cognitive exam
3. Answer questions about their medical history
4. Complete a few brief surveys about fatigue, balance, falls, freezing of gait, quality of life, and activities of daily living
5. Complete a 10-meter walk test
6. Wear the UG motion sensor (which detects FoG) on each ankle
7. Wear the PDVibe3 (which provides vibration) on each ankle
8. Walk five, 5-meter scenarios without vibration, and then again three more times with vibration therapy in a public setting on VCU campus. The five scenarios include:

   1. Walking through a narrow passage
   2. Walk and turn 540 degrees
   3. Walk toward a chair
   4. Walk while performing a verbal task
   5. Walk through a door before it closes

Participants will be able to take breaks at any time if they feel tired. Participants will be photographed and videotaped during the walking sessions, but faces will be blurred so that the recordings will not be identifiable.

Participation in this study can last up to 5 hours with several breaks. Approximately 20 individuals will participate in this study.

ELIGIBILITY:
Inclusion

* age >18 years,
* Parkinson's disease (PD) diagnosed by a movement disorder specialist using UK Brain Bank criteria,
* are able to walk independently or with a simple device (e.g., cane or walker), and
* are observed by the research team to have PD-related FoG in at least two of the five previously described common trigger scenarios (i.e., freezing upon gait initiation, walking through tight quarters, freezing when changing directions, approaching a visual target, dual tasking, and stressful, time sensitive situations such as entering an elevator before the doors close).

Exclusion

* individuals with known Parkinson plus syndrome,
* presence of dementia (Montreal Cognitive Assessment < 21),
* an additional disorder (not related to PD) impairing gait,
* history of implantable cardiac device or any other implanted electronic device except DBS,
* peripheral neuropathy (determined by use of tuning fork to check for ability to feel vibration),
* any condition that, in the opinion of the PI, would compromise participant safety, data integrity, or data interpretation,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vibration Therapy: 5-meter walk scenarios with vibration therapy
  UG motion sensor with PDVibe3: UG motion sensor (which detects FoG) on worn each ankle.
  PDVibe3 (which provides vibration) on worn each ankle
Period: Overall Study
Arm/Group | Vibration Therapy
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vibration Therapy
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Freezing of Gait (FoG) Episodes
Description: Participants will be videotaped during each walking task and the number of FoG episodes will be counted. Change in number of FoG episodes will be calculated by subtracting the average number of FoG episodes while experiencing vibration vs the number of episodes without vibration. For this test, the null hypothesis of no difference between the treatments versus the alternative hypothesis that the two groups differed.
Time Frame: Baseline to final walk task - up to 5 hours
Measure: Mean (Standard Error); unit: number of freezes
Arm/Group | Vibration Therapy
Number analyzed (Participants) | 12
number of freezes
  no vibration 540 degree turn/number of freezes | 3.75 (.765)
  vibration 540 degree turn/number of freezes | 5.17 (.765)
  no vibration narrow path/number of freezes | 4.0 (1.205)
  vibration narrow path/number of freezes | 3.63 (1.205)

2. Primary Outcome: Duration of Freezing of Gait (FoG) Episodes.
Description: Participants will be videotaped during each walking task and the duration of each FoG episodes will be calculated. Change in duration of FoG episodes will be calculated by subtracting the average duration of FoG episodes while experiencing vibration vs the average duration without vibration.
Time Frame: Baseline to final walk task - up to 5 hours
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Vibration Therapy
Number analyzed (Participants) | 12
minutes
  540 degree turn/no vibration/ total freezing time | 47.67 (12.06)
  540 degree turn/ vibration/ total freezing time | 52.14 (12.06)
  Narrow path/no vibration/ total freezing time | 34.565 (17.2)
  Narrow path/ vibration/ total freezing time | 43.505 (17.2)

ADVERSE EVENTS:
Time Frame: Baseline to final walk test, up to 5 hours
Arm/Group | Vibration Therapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibration Therapy (N=12)
Fall (Musculoskeletal and connective tissue disorders) | 10 (10) — This is an expected AE due to the population studied

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT04746846/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04746846/SAP_001.pdf
  • Informed Consent Form (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT04746846/ICF_002.pdf